CLINICAL TRIAL: NCT05923216
Title: Induction of Sustained Unresponsiveness to Sesame Using High- and Low-dose Sesame Oral Immunotherapy - Evaluation of Efficacy and Safety
Brief Title: Induction of Sustained Unresponsiveness to Sesame Using High- and Low-dose Sesame Oral Immunotherapy
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of Warsaw (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Sesame Protocol - SU
Record Dates: First submitted 2023-06-19; First posted 2023-06-28 (Actual); Last update posted 2025-01-31 (Actual); Status verified 2025-01

CONDITIONS: Food Allergy
Keywords: sesame; food allergy; sustained unresponsiveness; children
MeSH Terms: conditions — Food Hypersensitivity; SeSAME syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- High dose (Experimental): 20 patients Intervention: Dietary Supplement: High dose OIT
  Interventions: Dietary Supplement: High dose OIT
- Low dose (Active Comparator): 20 patients Intervention: Dietary Supplement: Low dose OIT
  Interventions: Dietary Supplement: Low dose OIT

INTERVENTIONS:
Dietary Supplement: High dose OIT — Patients will receive daily a high dose of the sesame paste (1200 mg sesame protein) mixed with well-tolerated fruit mousse or bread.
  Arms: High dose
Dietary Supplement: Low dose OIT — Patients will receive daily a low dose of the sesame paste (300 mg sesame protein) mixed with well-tolerated fruit mousse or bread.
  Arms: Low dose

SUMMARY:
This is an experimental, interventional study, following on from a clinical trial comparing the efficacy and safety of oral immunotherapy with low and high doses of sesame protein, in which patient desensitisation was achieved (High and Low Dose Oral Sesame Immunotherapy - Comparison of Efficacy and Safety, NCT05158413).

The aim of this study is to assess a sustained unresponsiveness (SU) to sesame protein after at least 8 months of previously assigned high- or low-dose sesame OIT, followed by 4-week-allergen avoidance, and verified by an open oral food challenge (OOFC).

DETAILED DESCRIPTION:
Oral immunotherapy is considered the most effective treatment for food allergy. There are two main goals of food immunotherapy: achievement of desensitisation and sustained unresponsiveness.

Desensitisation involves achieving temporary tolerance of the allergenic food by the patient only during regular intake of the allergen. The most desirable effect of immunotherapy is to achieve sustained unresponsiveness, i.e. to maintain the absence of adverse symptoms to a given allergen after specific immunotherapy has been discontinued for a defined period of time.

The study is a continuation of a clinical trial NCT05158413 which was designed to compare the efficacy and safety of oral immunotherapy (OIT) with low or high doses of sesame protein (300 or 1200 mg, respectively) in children with a confirmed diagnosis of sesame allergy. The participants of current study will be recruited from patients who have accomplished their per-protocol participation in previous trial.

Patients will receive the same maintenance dose of sesame allergen, which was used in previous trial (300 or 1200 mg, respectively), for 32 weeks (+/-2 weeks). Then, OIT will be discontinued for 4 weeks with strict sesame avoidance. Subsequently, an open oral food challenge (OOFC) will be performed to assess the achievement of sustained unresponsiveness.

ELIGIBILITY:
Inclusion Criteria:

* patients who have accomplished their per-protocol participation in trial NCT05158413.
* signed Informed Consent by parent/legal guardian and patient aged>16 years old
* patient's/caregiver's cooperation with researcher

Exclusion Criteria:

* severe asthma
* uncontrolled mild/moderate asthma: forced expiratory volume at one second (FEV1)<80% (under 5 percentile), FEV1/forced vital capacity (FEV)<75% (under 5 percentile), hospitalization due to asthma exacerbation within last 12 months
* current oral/sublingual/subcutaneous immunotherapy with another allergen
* eosinophilic esophagitis
* allergic reaction of 4th or higher grade according to the World Allergy Organisation Systemic Allergic Reaction Grading System during immunotherapy
* a history of severe recurrent anaphylaxis episodes
* chronic diseases requiring continous treatment, including heart disease, epilepsy, metabolic disease, diabetes
* medication:

  * oral, daily steroid therapy exceeding 1 month within the last 12 months
  * at least two courses of oral steroid therapy (at least 7 days) within the last 12 months
  * oral steroid therapy longer than 7 days within the last 3 months
  * biological treatment
  * the need to constantly take antihistamines
  * therapy with b-blockers, angiotensin converting enzyme (ACE) inhibitors, calcium channel inhibitors
* pregnancy
* no consent to participate in the study
* lack of patient cooperation

Ages: 4 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 40 (Estimated)
Dates: Start 2023-03-24 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
Sustained unresponsiveness to a sesame protein after discontinuing oral immunotherapy for 4 weeks. | Up to 9 months after starting maintenance phase
  Percentage of patients tolerating their maintenance dose of sesame protein after a 4-week break in immunotherapy
The highest tolerated dose of sesame protein after discontinuing oral immunotherapy for 4 weeks. | Up to 9 months after starting maintenance phase
  Sustained unresponsiveness assessed as the highest tolerated dose of sesame protein at oral food challenge.

SECONDARY OUTCOMES:
Adverse events | Up to 9 months after starting maintenance phase
  Number and severity of adverse events during OIT treatment and at OOFC will be assessed and compared between both groups.
Laboratory data | Up to 9 months after starting maintenance phase
  Change in sesame serum immunoglobulin E (IgE) level and immunoglobulin G4 (IgG4) level at different time points: before immunotherapy, at the end of the maintenance phase and after a 4-week break in immunotherapy, assessed for each individual and compared between groups.
Skin prick test (SPT) | Up to 9 months after starting maintenance phase
  Difference in wheal diameter in skin prick tests (SPT) assessed between groups at the respective time points: before immunotherapy, at the end of the maintenance phase and after a 4-week break in immunotherapy.
Tolerance of a single dose of 4000 mg of sesame protein | Up to 9 months after starting maintenance phase
  Percentage of patients tolerating a single dose of 4000 mg of sesame protein after a 4- week break in immunotherapy.

CONTACTS AND LOCATIONS:
Overall Officials: Katarzyna Grzela, PhD, MD, Study Chair — Medical University of Warsaw
Locations (1):
- Medical University of Warsaw, Warsaw, Poland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Sampson HA, Gerth van Wijk R, Bindslev-Jensen C, Sicherer S, Teuber SS, Burks AW, Dubois AE, Beyer K, Eigenmann PA, Spergel JM, Werfel T, Chinchilli VM. Standardizing double-blind, placebo-controlled oral food challenges: American Academy of Allergy, Asthma & Immunology-European Academy of Allergy and Clinical Immunology PRACTALL consensus report. J Allergy Clin Immunol. 2012 Dec;130(6):1260-74. doi: 10.1016/j.jaci.2012.10.017. No abstract available. PMID 23195525
- [Background] Pajno GB, Fernandez-Rivas M, Arasi S, Roberts G, Akdis CA, Alvaro-Lozano M, Beyer K, Bindslev-Jensen C, Burks W, Ebisawa M, Eigenmann P, Knol E, Nadeau KC, Poulsen LK, van Ree R, Santos AF, du Toit G, Dhami S, Nurmatov U, Boloh Y, Makela M, O'Mahony L, Papadopoulos N, Sackesen C, Agache I, Angier E, Halken S, Jutel M, Lau S, Pfaar O, Ryan D, Sturm G, Varga EM, van Wijk RG, Sheikh A, Muraro A; EAACI Allergen Immunotherapy Guidelines Group. EAACI Guidelines on allergen immunotherapy: IgE-mediated food allergy. Allergy. 2018 Apr;73(4):799-815. doi: 10.1111/all.13319. Epub 2017 Dec 5. PMID 29205393
- [Background] Adatia A, Clarke AE, Yanishevsky Y, Ben-Shoshan M. Sesame allergy: current perspectives. J Asthma Allergy. 2017 Apr 27;10:141-151. doi: 10.2147/JAA.S113612. eCollection 2017. PMID 28490893
- [Background] Burks AW, Sampson HA, Plaut M, Lack G, Akdis CA. Treatment for food allergy. J Allergy Clin Immunol. 2018 Jan;141(1):1-9. doi: 10.1016/j.jaci.2017.11.004. PMID 29307409
- [Background] Nachshon L, Goldberg MR, Levy MB, Appel MY, Epstein-Rigbi N, Lidholm J, Holmqvist M, Katz Y, Elizur A. Efficacy and Safety of Sesame Oral Immunotherapy-A Real-World, Single-Center Study. J Allergy Clin Immunol Pract. 2019 Nov-Dec;7(8):2775-2781.e2. doi: 10.1016/j.jaip.2019.05.031. Epub 2019 May 29. PMID 31150789
- [Background] Dalal I, Goldberg M, Katz Y. Sesame seed food allergy. Curr Allergy Asthma Rep. 2012 Aug;12(4):339-45. doi: 10.1007/s11882-012-0267-2. PMID 22610362